## Evaluation of Preventive (Stay Safe) Training Program of Child Abuse for Teachers and Children: A Randomized Controlled Trial from Multan City

Statistical Analysis Plan of the study

By

Zainab Noor Hussain
PSY-07
M.Phil. Applied Psychology

**Supervisor** 

Dr. Rizwana Amin



**Department of Applied Psychology** 

Bahauddin Zakariya University, Multan

Date: September 15, 2018

Statistical analysis

After collecting the data through questionnaires and completing the evaluation via SPSS

version 21.0, one way ANCOVAs is used for analysis as it clearly describes the effect of

intervention on students and teachers. There are sub scales of questionnaire and each sub scale

is being analyzed by one way ANCOVA for better understanding of the each aspect in regards

to intervention. Descriptive statistics of students and teachers are also explained in

the form of tables. Now, difference would be more easily assessable through this analysis.

**Ethical consideration** 

Before initiating the study, informed consent taken from teachers and parents of children to get

their willingness to participate in the study and also to get an idea about research. It also ensure

their confidentiality and privacy of the data which encourage them to participate more

confidently. As control group receive no training so it is necessary to inform them after

completing the research. Debriefing the research purpose and training ides to the control group

after completing the research study. It will be ensure that participant's rights would be

considered and prefer during the research study. All procedures and training methods will be

deliver to participants carefully to understand their feelings and emotions and also respect their

response.